CLINICAL TRIAL: NCT02905877
Title: The Pathophysiology of Functional Neurological Disorders
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 16/0275
Record Dates: First submitted 2016-09-02; First posted 2016-09-19 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Functional Neurological Disorders
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Functional neurological disorders: Initially especially patients diagnosed with a functional tremor.
  Interventions: Other: Behavioural study
- Organic neurological disorders.: Initially especially patients diagnosed with a an organic action tremor (e.g. essential tremor or dystonic tremor).
  Interventions: Other: Behavioural study
- Healthy control: Healthy age matched controls
  Interventions: Other: Behavioural study

INTERVENTIONS:
Other: Behavioural study — reaching studies and other behavioural studies.

SUMMARY:
Functional disorders, also called psychogenic or psychosomatic are very common, disabling and their costs to society are immense.

Functional movement disorders are abnormal, involuntary movements, that are illogical in terms of classic neurology. Intriguingly, they typically manifest when patients pay attention to them and disappear with distraction.

The investigators aim to further the understanding of the pathophysiological mechanisms underlying functional neurological disorders in order to improve treatment. In particular they aim to understand the effect of attention on movement in general, on functional neurological mechanisms and on the sense of agency (of subjective control) over a movement.

Patients with a functional neurological disorder, patients with an organic neurological disorder and healthy participants will perform simple tasks, such as reaching to a target, while additional tasks will manipulate their attention. The effects of these attentional manipulations will be analysed on several levels: movement performance, analysed by the kinematics and electromyography (EMG),and psychophysical measures, such as the sense of agency.

If the hypothesis turns out to be true, then changing the attentional focus could be used as a treatment in functional neurological disorders.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit three groups of participants:

  1. functional neurological disorders, e.g. functional tremor: diagnosed by a neurologist.
  2. organic counterpart of the functional neurological disorders, e.g. in the case of functional tremor, the organic counterpart would be organic tremor: presence of an organic tremor according to internationally recognised guidelines and diagnosed by a neurologist.
  3. healthy age-matched controls.

Exclusion Criteria

* Healthy Participants: Major neurological disorder.

All groups:

1. Age under 18 or over 80
2. Significant impairment in ability to give informed consent for study procedures due to significant cognitive impairment and/or inability to understand study literature,
3. very severe tremor
4. moderate or severe cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: see below under inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Tremor severity, assessed by kinematics, under different attentional conditions | 1 year

SECONDARY OUTCOMES:
Sense of agency, assessed by intentional binding, under different attentional conditions | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Neurology, University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No